CLINICAL TRIAL: NCT06687811
Title: The Effects of Preoperative Carbohydrate Loading on Perioperative Blood Glucose Levels and Insulin Resistance in Type 2 Diabetes Mellitus Patients Undergoing Elective Surgery
Brief Title: Carbohydrate Loading in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aries Perdana, Staff of Departement of Anesthesiology and Intensive Care, Division of Cardiac Anesthesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IndonesiaUAnes093
Record Dates: First submitted 2024-11-10; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Carbohydrate loading; Type 2 Diabetes Mellitus; Perioperative blood glucose; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbohydrate loading (CHO) group (Active Comparator): Patient received preoperative carbohydrate loading of 200 ml Maltodextrin 12.5%, given 2 hours before the operation
  Interventions: Other: preoperative carbohydrate loading
- Control (Placebo Comparator): Patient received preoperative regular drinking water of 200 ml with zero-calorie sweetener, given 2 hours before the operation
  Interventions: Other: Placebo

INTERVENTIONS:
Other: preoperative carbohydrate loading — Patients receive 200 ml drink containing Maltodextrin 12.5%, 2 hours prior to surgery
  Other Names: CHO
  Arms: Carbohydrate loading (CHO) group
Other: Placebo — Patients receive 200 ml regular drinking water with zero-calorie sweetener, 2 hours prior to surgery
  Other Names: Control
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn the effects of preoperative carbohydrate loading on perioperative blood glucose levels and insulin resistance in type 2 diabetes mellitus undergo elective surgery. The main questions it aims to answer are:

* Does carbohydrate loading affects perioperative blood glucose and insulin resistance in type 2 diabetes mellitus patients undergo surgery?
* How are the incident of perioperative hyperglycemia and hypoglycemia between subjects who receive placebo compared with subjects who receive carbohydrate loading
* How are the hyperglycemia-related complications comparison between two groups?

Researchers will compare the carbohydrate loading intervention to placebo (regular drinking water with zero-calorie sweetener) to see the effects of carbohydrate loading to blood glucose levels and insulin resistance (by HOMA-IR value)

Participants will:

* randomized to carbohydrate loading (CHO) group or placebo
* checked for preoperative, intraoperative, postoperative blood glucose, and preoperative and postoperative insulin level
* evaluated for any hyperglycaemia-related complications

ELIGIBILITY:
Inclusion Criteria:

* Controlled type 2 diabetes mellitus with any treatment
* BMI <30 kg/m2
* Non-major elective surgery

Exclusion Criteria:

* Subject refusal
* Geriatric patients with frailty score >4
* Subjects with critical illness
* Subjects received steroid treatment
* Subjects received total parenteral nutrition
* Subjects with intestinal obstruction
* Subjects with impaired liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Perioperative Blood Glucose Level | Preoperative (before intervention), 1 hour intraoperative, 30 minutes postoperative, 1 day postoperative
  Blood glucose sampled from vein and capillary, measured in mg/dL
Insulin Resistance | preoperative and 30 minutes postoperative
  Calculated using Homeostasis Model Assessment Insulin Resistance (HOMA-IR), obtained from measured fasting insulin (μU/ml) × fasting glucose (mmol/l) / 22.5

SECONDARY OUTCOMES:
Abnormal blood glucose incidence | Preoperative, 1 hour intraoperative, 30 minutes postoperative, 1 day postoperative
  Blood glucose level below 60 mg/dL (hypoglycaemia) or above 200 mg/dL (hyperglycaemia)
Complications | Up to 1 week postoperative or discharged from hospital stay
  Hyperglycaemia-related complications, such as surgical site infection, aspiration, prolonged length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Cipto Mangunkusumo, Central Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to erika.sasha@ui.ac.id. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years after publication at a third party website (link in process will be updated to be included)

REFERENCES:
- [Background] Ljungqvist O, Nygren J, Thorell A. Modulation of post-operative insulin resistance by pre-operative carbohydrate loading. Proc Nutr Soc. 2002 Aug;61(3):329-36. doi: 10.1079/PNS2002168. PMID 12230794
- [Background] Weledji EP, Njong SN, Chichom A, Verla V, Assob JC, Ngowe MN. The effects of preoperative carbohydrate loading on the metabolic response to surgery in a low resource setting. Int J Surg Open. 2017;8:18-23.
- [Background] Robinson KN, Cassady BA, Hegazi RA, Wischmeyer PE. Preoperative carbohydrate loading in surgical patients with type 2 diabetes: Are concerns supported by data? Clin Nutr ESPEN. 2021 Oct;45:1-8. doi: 10.1016/j.clnesp.2021.08.023. Epub 2021 Sep 3. PMID 34620304
- [Background] Pogatschnik C, Steiger E. Review of Preoperative Carbohydrate Loading. Nutr Clin Pract. 2015 Oct;30(5):660-4. doi: 10.1177/0884533615594013. Epub 2015 Jul 21. PMID 26197803
- [Background] Bilku DK, Dennison AR, Hall TC, Metcalfe MS, Garcea G. Role of preoperative carbohydrate loading: a systematic review. Ann R Coll Surg Engl. 2014 Jan;96(1):15-22. doi: 10.1308/003588414X13824511650614. PMID 24417824
- [Background] Lin MW, Chen CI, Cheng TT, Huang CC, Tsai JW, Feng GM, Hwang TZ, Lam CF. Prolonged preoperative fasting induces postoperative insulin resistance by ER-stress mediated Glut4 down-regulation in skeletal muscles. Int J Med Sci. 2021 Jan 11;18(5):1189-1197. doi: 10.7150/ijms.52701. eCollection 2021. PMID 33526980
- [Background] Elias KM, Stone AB, McGinigle K, Tankou JI, Scott MJ, Fawcett WJ, Demartines N, Lobo DN, Ljungqvist O, Urman RD; ERAS(R) Society and ERAS(R) USA. The Reporting on ERAS Compliance, Outcomes, and Elements Research (RECOvER) Checklist: A Joint Statement by the ERAS(R) and ERAS(R) USA Societies. World J Surg. 2019 Jan;43(1):1-8. doi: 10.1007/s00268-018-4753-0. PMID 30116862
- [Background] Soop M, Nygren J, Myrenfors P, Thorell A, Ljungqvist O. Preoperative oral carbohydrate treatment attenuates immediate postoperative insulin resistance. Am J Physiol Endocrinol Metab. 2001 Apr;280(4):E576-83. doi: 10.1152/ajpendo.2001.280.4.E576. PMID 11254464
- [Background] Thorell A, Nygren J, Hirshman MF, Hayashi T, Nair KS, Horton ES, Goodyear LJ, Ljungqvist O. Surgery-induced insulin resistance in human patients: relation to glucose transport and utilization. Am J Physiol. 1999 Apr;276(4):E754-61. doi: 10.1152/ajpendo.1999.276.4.E754. PMID 10198313
- [Background] Gutch M, Kumar S, Razi SM, Gupta KK, Gupta A. Assessment of insulin sensitivity/resistance. Indian J Endocrinol Metab. 2015 Jan-Feb;19(1):160-4. doi: 10.4103/2230-8210.146874. PMID 25593845
- [Background] Duggan EW, Carlson K, Umpierrez GE. Perioperative Hyperglycemia Management: An Update. Anesthesiology. 2017 Mar;126(3):547-560. doi: 10.1097/ALN.0000000000001515. PMID 28121636
- [Background] Gillis C, Carli F. Promoting Perioperative Metabolic and Nutritional Care. Anesthesiology. 2015 Dec;123(6):1455-72. doi: 10.1097/ALN.0000000000000795. PMID 26248016
- [Background] Makuuchi R, Sugisawa N, Kaji S, Hikage M, Tokunaga M, Tanizawa Y, Bando E, Kawamura T, Terashima M. Enhanced recovery after surgery for gastric cancer and an assessment of preoperative carbohydrate loading. Eur J Surg Oncol. 2017 Jan;43(1):210-217. doi: 10.1016/j.ejso.2016.07.140. Epub 2016 Aug 10. PMID 27554250
- [Background] Albalawi Z, Laffin M, Gramlich L, Senior P, McAlister FA. Enhanced Recovery After Surgery (ERAS(R)) in Individuals with Diabetes: A Systematic Review. World J Surg. 2017 Aug;41(8):1927-1934. doi: 10.1007/s00268-017-3982-y. PMID 28321553
- [Background] Gustafsson UO, Nygren J, Thorell A, Soop M, Hellstrom PM, Ljungqvist O, Hagstrom-Toft E. Pre-operative carbohydrate loading may be used in type 2 diabetes patients. Acta Anaesthesiol Scand. 2008 Aug;52(7):946-51. doi: 10.1111/j.1399-6576.2008.01599.x. Epub 2008 Mar 7. PMID 18331374
- [Background] Awad S, Varadhan KK, Ljungqvist O, Lobo DN. A meta-analysis of randomised controlled trials on preoperative oral carbohydrate treatment in elective surgery. Clin Nutr. 2013 Feb;32(1):34-44. doi: 10.1016/j.clnu.2012.10.011. Epub 2012 Nov 7. PMID 23200124
- [Background] Alimena S, Falzone M, Feltmate CM, Prescott K, Contrino Slattery L, Elias K. Perioperative glycemic measures among non-fasting gynecologic oncology patients receiving carbohydrate loading in an enhanced recovery after surgery (ERAS) protocol. Int J Gynecol Cancer. 2020 Apr;30(4):533-540. doi: 10.1136/ijgc-2019-000991. Epub 2020 Feb 26. PMID 32107317
- [Background] Talutis SD, Lee SY, Cheng D, Rosenkranz P, Alexanian SM, McAneny D. The impact of preoperative carbohydrate loading on patients with type II diabetes in an enhanced recovery after surgery protocol. Am J Surg. 2020 Oct;220(4):999-1003. doi: 10.1016/j.amjsurg.2020.03.032. Epub 2020 Mar 30. PMID 32252984
- [Background] Gachabayov M, Senagore AJ, Abbas SK, Yelika SB, You K, Bergamaschi R. Perioperative hyperglycemia: an unmet need within a surgical site infection bundle. Tech Coloproctol. 2018 Mar;22(3):201-207. doi: 10.1007/s10151-018-1769-2. Epub 2018 Mar 6. PMID 29512047